CLINICAL TRIAL: NCT01716182
Title: RAMP Study: A Prospective Randomized Study Comparing Two Lumbar Fusion Procedures
Brief Title: RAMP Study: A Study Comparing Two Lumbar Fusion Procedures
Acronym: RAMP
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: Baxano Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-0018
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Stenosis; Spondylolisthesis; Degenerative Disc Disease
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- transacral lumbar interbody fusion procedure
- transforaminal lumbar interbody fusion procedure (TLIF)

SUMMARY:
This is a post-marketing, on-label Efficacy, Effectiveness and Safety Study designed in a Multicenter, Randomized, Prospective format. This study compares two spinal fusion procedures, Transacral Interbody Fusion and Transforaminal Lumbar Interbody Fusion (TLIF). Enrollment period will be approximately 12-18 months; each Principal Investigator/Study Center will be expected to enroll up to 20 subjects. The protocol requires approximately 7 subject visits to the study center from screening through the final follow-up visit.

DETAILED DESCRIPTION:
Study Treatment Arms:

The transacral lumbar interbody fusion (including 1L+ and 2L+) is a minimally invasive technique that uses a transacral approach to achieve fusion at the L5-S1 or L4-L5-S1 spinal levels. The transforaminal lumbar interbody fusion (TLIF) is performed by using a posterior unilateral or bilateral incision in which the lumbar spine is accessed. Both study procedures are approved for use and conform to US regulatory requirements. The study employs these procedures and devices for uses that are consistent with their 510(k), legally cleared, labeling.

Study Design, Objective:

The study objective is to demonstrate non-inferiority between the transacral lumbar interbody fusion procedure and the transforaminal lumbar interbody fusion procedure (TLIF) by meeting the primary and secondary study endpoints as listed below.

Study design, Endpoints:

Primary Endpoint:

Efficacy: Fusion of the targeted vertebral bodies (L4-L5 or L5-S1) by 24 months as determined by Central Radiographic Reviewer's interpretation of high resolution Computed Tomography (CT) scan.

Secondary Endpoints:

Safety: Incidence of major device-related adverse events and/or failures by 24 months, defined as those requiring revision surgery or a secondary operation, or events resulting in permanent disability or death.

Clinical Effectiveness: A 20% decrease in back pain compared to baseline by 24 months as measured by the Visual Analog Scale (VAS) score.

Clinical Effectiveness: A 20% decrease in disability compared to baseline by 24 months as measured by the Oswestry Disability Index (ODI).

Study Design, Enrollment and Analyses:

Approximately 200 subjects will be enrolled in this study and will receive one of two study treatments in the study. The enrollment period is expected to last approximately 18 months, with a 24 month follow up period. Approximately 15-20 sites will participate, and Investigators must be proficient in both of the lumbar fusion procedures.

Analyses:

Eight evaluations: Pre-Operative, Operative, Discharge, and at 1, 3, 6, 12, and 24 Months.

Safety and efficacy analyses will be performed at all follow-up points during the study as well as a final analysis when all subjects have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject that is eligible for both study procedures only at the L4-L5-S1 or L5-S1 levels with bilateral pedicle screws;
* The subject has a diagnosis of one or more of the following conditions at the L4-L5-S1 or L5-S1 levels:

  * Spinal stenosis;
  * Spondylolisthesis;
  * Degenerative Disc Disease (DDD) defined as back pain and/or radicular pain with degeneration of the disc as confirmed by history, physical examination and radiographic studies, either by CT, MRI, plain film, myelography, or discography;
* Adult 18 years of age or older;
* The subject has undergone at least 6 consecutive months of Conservative Care Therapy(ies);
* The subject is able and willing to give written informed consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

* Coagulopathy;
* Bowel disease (e.g. Crohn's, ulcerative colitis);
* Severe scoliosis (curves > 60°);
* Sacral agenesis;
* Spondylolisthesis greater than Grade 1 at the L4-L5-S1 levels, or greater than Grade 2 at the L5-S1 level;
* Spinal tumor (or history of sacral tumor);
* History of fracture at L4, L5 and/or S1 vertebral bodies;
* The subject has undergone a prior fusion procedure of the lumbar spine;
* Osteoporosis; or, if the subject is at high risk for development of osteoporosis, further screening to be conducted at Investigator's discretion;
* Per the Investigator, body weight is exclusionary only if concomitant medical issues are present that preclude the subject from being a candidate for spinal surgery; The subject is a current cigarette smoker;
* For women of childbearing potential, pregnancy at the time of enrollment, or planning to become pregnant during the course of the study;
* The subject has a history of substance abuse (illegal drugs, prescription drugs, or alcohol) that, in the Investigator's opinion, may interfere with protocol assessments and/or the subject's ability to comply with the protocol;
* Per the Investigator, the subject is in poor general health or undergoing any concurrent disease process that would place the subject in excessive risk to surgery (e.g. significant circulatory problems, cardiac disease, history of bowel surgery);
* The subject is participating in another spine study, which, in the opinion of the Investigator, could skew results;
* The subject is involved in litigation related to their back condition;
* The subject is contraindicated to receive either study procedure;
* The subject is contraindicated to receive bilateral pedicle screws;
* The subject has a history of allergy to any component of the devices or biologic material to be implanted in either procedure;
* The subject is a prisoner, transient, or an illegal alien.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be eligible to participate in this study, the subject must meet all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 24 months post-operative
  Efficacy: Fusion of the targeted vertebral bodies (L4-L5-S1 or L5-S1) will be assessed individually at 24 months as determined by Central Radiographic Reviewer's (orthopedic surgeon) interpretation of high resolution Computed Tomography (CT) Scan.

CONTACTS AND LOCATIONS:
Overall Officials: David Hart, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (11):
- United States (11):
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana Spine Group, Carmel, Indiana
  - Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana
  - LSU Health Sciences Center, Department of Neurosurgery, New Orleans, Louisiana
  - UMass Medical Center, Department of Neurosurgery, Worcester, Massachusetts
  - Cary Orthopaedic Spine Specialists, Cary, North Carolina
  - Mayfield Clinic/University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Brazos Spine, College Station, Texas
  - Danville Orthopedic Clinic, Inc., Danville, Virginia